CLINICAL TRIAL: NCT01089244
Title: Molecular Correlates and Clinical Significance of Positron Emission Tomography With FET-PET in Combination With Perfusion-weighted Magnetic Resonance Imaging (PWI) in Patients With Low Grade Gliomas
Brief Title: FET-PET for Diagnosis and Monitoring in Patients With Low Grade Glioma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Bogdana Suchorska, PI, Ludwig-Maximilians - University of Munich
Other Study IDs: GGN-CP4
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Astrocytoma; Oligoastrocytoma; Oligodendroglioma
Keywords: Low grade glioma; Astrocytoma; Molecular imaging; FET PET; Therapy monitoring; Temodar
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — High molecular wight DNA and RNA speciments for MGMT promoter methylation, IDH1/IDH2 and p53 mutation, LOH 1p and 19q analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients with a suspected WHO II low grade glioma, disease progression within
  1 year
- Group B: Patients with a suspected WHO II low grade glioma, progression free within 1 year

SUMMARY:
The aim of the study is to compare the two imaging modalities perfusion weighted MR-imaging and FET-PET in their ability to provide an accurate histological evaluation of low grade glioma and to reveal focal abnormalities within a homogeneously appearing tumor. Additionally, therapeutic effects should be assessed during a time period of two years.

ELIGIBILITY:
Inclusion Criteria:

* neuroradiologically suspected low grade glioma (Astrocytoma WHOI-II, Oligodendroglioma WHO II, Oligoastrocytoma WHO II)
* histological verification will be obtained either by microsurgery or by stereotactic biopsy
* patients older than 18 years
* Karnofsky Performance Score >=70
* pregnant or nursing female patients will not be included in this study

Exclusion Criteria:

* patients in whom informed consent cannot be obtained due to organic brain syndrome or insufficient language skills
* patients who cannot lie quiet for a time period of app. two hours during the FET-PEt scan
* medical history of a metastatic brain disease
* patients in whom an MRI scan cannot be performed due to claustrophobia metallic protheses or pacemakers etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a suspected referred to a Neurosurgical Department in order to provide a diagnosis and therapy
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2008-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months

SECONDARY OUTCOMES:
Progression Free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C. Tonn, Prof. Dr., Principal Investigator — Department of Neurosurgery, LMU Munich
Locations (2):
- Germany (2):
  - University Hospital Munich, Department of Neurosurgery, Munich, Bavaria
  - University Hospital, Duesseldorf, Düsseldorf, North Rhine-Westphalia